CLINICAL TRIAL: NCT06627894
Title: Attenuating DEPression With Internet CBT to Slow Cognitive Decline in Older ICU Survivors(ADEPT-ICU)
Acronym: ADEPT-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Babar Khan, MD, MS, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22761; 1R01AG084754-01A1 (NIH)
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Depression; Cognitive Decline
Keywords: Depression; Cognition
MeSH Terms: conditions — Depression; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Internet based CBT-D vs Active Control
Who Masked: Investigator, Outcomes Assessor
Masking Description: The unblinded study coordinator is aware of randomization. The investigator and study team members responsible for the delivery of the intervention will be unblinded.
  The study team staff performing outcomes assessments and the investigators overseeing this process will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Internet Cognitive-Behavioral Therapy (CBT) for Depression (Experimental): Participants will complete nine 45-minute sessions of an internet CBT for depression called Good Days Ahead (GDA; MindStreet, Inc.) with 20 minutes of therapist assistance per session on the phone over six months.
  Interventions: Behavioral: Therapist-Assisted Internet Cognitive-Behavioral Therapy for Depression
- Active Control - Depression Education, Symptom Monitoring, and Usual Care (Active Comparator): Participants will review nine 45-minute segments of depression education material on their own with 20 minutes of therapist assistance per segment on the phone over six months. They will also have access to and could receive current depression care in the targeted healthcare systems.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Therapist-Assisted Internet Cognitive-Behavioral Therapy for Depression — Good Days Ahead (MindStreet, Inc.)
  Arms: Intervention - Internet Cognitive-Behavioral Therapy (CBT) for Depression
Behavioral: Active Control — Depression education, symptom monitoring, and standard depression care
  Arms: Active Control - Depression Education, Symptom Monitoring, and Usual Care

SUMMARY:
Depression affects one-third of intensive care unit (ICU) survivors and represents a potentially modifiable target to slow cognitive decline and reduce the risk of Alzheimer's disease and related dementias (ADRD). Our multi-PI team proposes a two-arm RCT called ADEPT-ICU (Attenuating DEPression with Internet CBT to Slow Cognitive Decline in Older ICU Survivors), which will test the efficacy of an internet CBT intervention called Good Days Ahead (GDA) to reduce the burden of subjective cognitive decline (SCD) in older ICU survivors with moderate to severe depressive symptoms after ICU hospitalization.

DETAILED DESCRIPTION:
Alzheimer's disease and related dementias (ADRD) affect 47 million people worldwide with an annual global cost of $818 billion. The risk of developing ADRD is disproportionately borne by older adults with multiple chronic conditions from underrepresented racial and ethnic groups (URGs). One such high risk group is older survivors of critical illness who were admitted to the intensive care units (ICUs). Nearly half of ICU survivors experience subjective cognitive decline(SCD), i.e., perceived decline in memory and thinking even with normal objective cognitive data. With over 5 million adult ICU admissions in the US each year, an intervention reducing SCD in older ICU survivors could significantly prevent or lower the incidence of ADRD. Thus, there is an urgent need for an inclusive randomized controlled trial (RCT) to rigorously test whether a novel, accessible, and scalable intervention can reduce SCD in a diverse cohort of older ICU survivors. One potential target for such interventions is post-ICU depression, which affects about one-third of ICU survivors. To date, there are no large scale RCTs which have rigorously tested whether depression focused psychotherapies, such as cognitive behavioral therapy (CBT), reduce SCD in a diverse cohort of older ICU survivors with depression.

We propose a two-arm, randomized, parallel-group, assessor-blinded clinical trial to evaluate the efficacy of internet CBT for depression compared to an active control in reducing SCD and slowing cognitive decline in older ICU survivors with post-ICU depression. The total duration of the intervention will be 6 months from randomization.

ELIGIBILITY:
Inclusion Criteria

1. 50 years of age and older
2. Admitted to the intensive care for greater > 48 hours
3. Able to understand and provide informed consent
4. Elevated depressive symptoms, defined as Screening PHQ-9 or PHQ-8 ≥ 10 or Screening PHQ-9 or PHQ-8 = 5-9 with the presence a core symptom of anhedonia (PHQ-9 or PHQ-8 Item 1) or depressed mood (PHQ-9 or PHQ-8 Item 2)
5. Willing to participate in cognitive testing
6. Access to a telephone
7. Discharge to home or an independent or assisted living facility
8. Response is a 1,2, or 3 on PHQ-9 or PHQ-8 item 7, answered yes to "Have you experienced a change in your memory or other aspect of thinking in the past 1 to 3 years?", or score in the 25% percentile or lower on the Montreal Cognitive Assessment (MOCA) based on normative data which account for age, gender, race, ethnicity and education.

Exclusion Criteria:

1. Diagnosis of dementia or neurodegenerative disease (e.g. Alzheimer's disease, vascular dementia as per EHR and IQCODE, or Parkinson's disease) or on anti-dementia medications prior to ICU stay
2. Diagnosis of severe mental illness (bipolar disorder, schizophrenia, schizoaffective) as per EHR and screening questions
3. Persistent psychotic symptoms after ICU stay which would interfere with successful completion of intervention
4. Recent or recurrent alcohol or substance use disorder as per HER and Drug Abuse Screening Test
5. Life expectancy less than 1 year (e.g. terminal cancer diagnosis, discharged on hospice)
6. Ischemic or hemorrhagic stroke, traumatic brain injury, or undergoing neurosurgery prior, during or after ICU stay
7. Uncorrected visual or auditory impairment including legal blindness or deaf
8. Status post tracheostomy and not able to communicate
9. Incarcerated or on parole after ICU stay

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Subjective Cognitive Decline | Measured at 6-month and 12-month follow-up.
  The primary outcome will be subjective cognitive decline (SCD), measured using the Cognitive Change Index self-report version (CCI-SR).

SECONDARY OUTCOMES:
Cognition status | Measured at 6-month and 12-month follow-up.
  Repeatable Battery for Assessment of Neuropsychological Status (RBANS)
Quality of Life physical and mental component status | Measured at 6-month and 12-month follow-up.
  Medical Outcome Study Short Form (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Babar Khan, MD, MS, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana